CLINICAL TRIAL: NCT02568514
Title: Study of the Effect on Clinical Outcomes Using Secure Text Messaging
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 823096
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Congestive Heart Failure; Diabetes; Renal Failure; Copd
Keywords: mhealth; text messaging; secure text messaging; communication
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus; Renal Insufficiency; Pulmonary Disease, Chronic Obstructive; Communication

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Patients admitted to hospital floors without any other intervention.
- Secure text messaging (Experimental): Patients admitted to hospital floors on which physicians and other staff are able to communicate with each other (not to the patient) using mobile secure text messaging.
  Interventions: Device: Secure text messaging

INTERVENTIONS:
Device: Secure text messaging — A smartphone and web application that allows physicians and other health care professionals to communicate to each other by secure text message
  Arms: Secure text messaging

SUMMARY:
In this study, the investigators will conduct a randomized, controlled trial to evaluate the impact of offering mobile secure text messaging on clinical outcomes.

DETAILED DESCRIPTION:
Inpatient health care providers such as physicians and nurses spend up to one-third of their time communicating with other health care providers. Many of these communications have shifted mediums from handwritten notes and face-to-face conversations to phone calls and paging systems. More recently the rapid adoption of smartphones has led to the use of mobile-enabled technologies using smartphones such as text messaging and email. While these technologies may offer ease and fit better within the clinical workflow, they often send patient information through unsecure cellular or internet connections. Mobile secure text messaging may address these issues by encrypting data and allowing for asynchronous or synchronous communication between individual providers or groups of providers. In this study, the investigators will conduct a randomized, controlled trial to evaluate the impact of offering mobile secure text messaging on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Admission to one of the hospital floors or services in the study at the Hospital of the University of Pennsylvania

Exclusion Criteria:

* Discharges against medical advice
* Discharges to hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change in length of stay | 6 months
  Change in inpatient length of stay from baseline to 6 months
Change in 30 day hospital readmissions | 6 months
  Change in 30 day hospital readmissions from baseline to 6 months
Change in inpatient mortality | 6 months
  Change in inpatient mortality from baseline to 6 months

SECONDARY OUTCOMES:
Change in Hospital Consumer Assessment of Healthcare Providers and Systems (HCAPs) scores | 6 months
  Change in HCAP scores from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States